CLINICAL TRIAL: NCT07066124
Title: The Effect of Progressive Relaxation Exercises on Sleep Quality and Quality of Life of Pregnant Women
Brief Title: Do Progressive Relaxation Exercises Affect the Sleep and Quality of Life of Pregnant Women?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Esra Bozhan Tayhan, Research Assistant, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: -Es-Ra!!Cbu
Record Dates: First submitted 2025-04-10; First posted 2025-07-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Sleep Quality; Quality of Life
Keywords: Pregnancy; progressive relaxation exercise; sleep quality; quality of life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises Group (Experimental): PRE training was given to the pregnant women in the intervention group and their practice was provided for six weeks.
  Interventions: Behavioral: Progressive Relaxation Exercises training was given to the pregnant women in the intervention group and their practice was provided for six weeks.
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercises training was given to the pregnant women in the intervention group and their practice was provided for six weeks. — Progressive Relaxation Exercises training was given to the pregnant women in the intervention group and their practice was provided for six weeks. After the first encounter, Pittsburgh Sleep Quality Index and Quality of Life Scale were re-administered to the pregnant women in the third and sixth weeks to evaluate their sleep and quality of life.
  Arms: Exercises Group

SUMMARY:
Aim: To examine the effects of progressive relaxation exercises (PRE) applied to pregnant women on sleep and life quality of pregnant women.

Methods: The research was carried out as a randomized controlled experimental study with pregnant women who applied to obstetrics clinics of a hospital. The research sample consisted of 66 pregnant women in the intervention and control groups. 'Pregnant Identification Form', 'Pittsburgh Sleep Quality Index' and Quality of Life Scale were applied to the pregnant women, and progressive relaxation exercises training was given to the pregnant women in the intervention group by randomization, and their practice was provided for six weeks. The control group received routine care. After the first encounter, Pittsburgh Sleep Quality Index and Quality of Life Scale were re-administered to the pregnant women in the third and sixth weeks to evaluate their sleep and quality of life. The data obtained were evaluated using the SPSS 15.0 program using descriptive statistics, chi-square cross tables, Independent simple t test, Repeated Measures test.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35
* Literate
* Primiparous
* Between 30-32 weeks of gestation
* Owns a smartphone to listen to the music included in the exercise content
* Willing to participate in the study

Exclusion Criteria:

* Having a high-risk pregnancy (gestational diabetes, eclampsia, preeclampsia, threat of preterm birth, premature rupture of membranes, placental anomalies, etc.)
* Conceiving through IVF (In Vitro Fertilization) treatment
* Having a maternal physical anomaly
* Experiencing communication difficulties or mental inadequacy
* No history of mental illness in medical history
* Detection of fetal anomalies during pregnancy
* Development of any disease/complication during pregnancy
* Not regularly practicing PRE
* Not wishing to continue with the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Progressive relaxation exercises have a positive effect on the sleep quality of pregnant women. | six weeks
  Progressive Relaxation Exercises (PRE) are breathing and stretching technique that helps relax nerves and muscles from hand to foot and, reduces sympathetic nervous system activity by stimulating the parasympathetic nervous system. It is thought that at the end of the PGE training given to pregnant women, learning PGE and applying it for six weeks will reduce the sleep problems that increase especially in the third trimester and thus increase their sleep and life quality. The PSQI evaluates sleep quality over the past month and consists of a total of 24 questions. The self-report questions cover various factors related to sleep quality, including estimates of sleep duration, sleep latency, and the frequency and severity of specific sleep-related issues. The scoring includes 18 items, grouped into 7 component scores. The sum of the component scores yields the total PSQI score, which ranges from 0 to 21. A total score greater than 5 indicates poor sleep quality.

SECONDARY OUTCOMES:
Progressive relaxation exercises have a positive effect on the quality of life of pregnant women. | six weeks
  The SF-12 encompasses two different dimensions: Physical Component Summary Score (PCSS) and Mental Component Summary Score (MCSS). Unlike the total score calculated for the SF-36, it is not used for the SF-12. In calculating the scale, the physical standardization values and mental standardization values for the answers given by individuals are added separately. Subsequently, for the 12 questions, 56.57706 is added to the physical standardization total to derive the physical components summary, and 60.75781 is added to the mental standardization total to derive the mental components summary. Both PCSS-12 and MCSS-12 scores range from 0 to 100, with higher scores representing better health. High scores indicate good health status. The Cronbach's alpha coefficients for the scale were found to be 0.73 for PCSS-12 and 0.72 for MCSS-12. In this study, the Cronbach's alpha coefficients were 0.69 for PCSS-12 and 0.71 for MCSS-12.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar Üniversitesi Sağlık Bilimleri Fakültesi, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No